CLINICAL TRIAL: NCT06474286
Title: A Pilot Study to Assess the Effect of Prucalopride on Cognitive Functioning in Patients With Schizophrenia
Brief Title: Prucalopride for Cognitive Functioning in Schizophrenia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH); K S Hegde Medical Academy (Unknown)
Responsible Party: Principal Investigator, Vishwajit Nimgaonkar, MD PhD, Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY23010044; D43TW009114 (NIH)
Record Dates: First submitted 2024-06-18; First posted 2024-06-25 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; neurocognitive impairment; cognitive deficits; Prucalopride
MeSH Terms: conditions — Schizophrenia; Cognition Disorders | interventions — prucalopride; Serotonin 5-HT4 Receptor Agonists

STUDY DESIGN:
Intervention Model Description: An open label, pilot study, interventional study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tab. Prucalopride (Experimental): The study drug Tab. Prucalopride 1 mg (30 tablets) will be dispensed to the participant. They will be explained to take one tablet of 1 mg Prucalopride per oral in the morning.
  Interventions: Drug: Prucalopride 1 MG

INTERVENTIONS:
Drug: Prucalopride 1 MG — The study drug Tab. Prucalopride 1 mg (30 tablets) will be dispensed to the participant. The drug will be procured at the local site manufactured in India only.They will be explained to take one tablet of 1 mg Prucalopride per oral in the morning. The participants will continue their antipsychotic regimen as per orders of their consultant and will continue to purchase their psychiatric medications as earlier. At the end of week 1, participants will be assessed for side effects via telephonic conversation.
  Other Names: 5HT4 receptor agonist

SUMMARY:
A core component of schizophrenia is neurocognitive impairment. The cognitive deficits are prominently seen in memory, attention, working memory, problem solving, processing speed and social cognition. Atypical antipsychotics continue to be the mainstay of treatment in schizophrenia.

Promising areas for future research include search for new compounds for cognition enhancement. Prucalopride, a highly selective 5HT4 receptor agonist is a potential drug and its effect on cognition in patients with schizophrenia needs to be studied.

An open label, pilot study involving 34 patients with schizophrenia diagnosed as per DSM 5 criteria. The participants will receive Tab. Prucalopride one milligram (1 mg) for a duration of four weeks along with their existing treatment regimen with antipsychotics.

Assessments includes PANSS and BACS at baseline and at the end of 4 weeks. The effect of prucalopride on cognitive functioning in patients with schizophrenia is studied.

DETAILED DESCRIPTION:
Prucalopride acts as a high affinity, high selective 5-hydroxy tryptamine receptor agonist. It is a gastrointestinal prokinetic drug predominantly used for constipation. In this study, the effect of prucalopride on cognitive functioning in schizophrenia is studied.

Participants who are diagnosed with schizophrenia, attending consultation at the outpatient department (OPD) of Psychiatry at K.S. Hegde Hospital and Nitte Rural Medical and Psychiatry Centre will be invited to participate in the study through their treating consultant. Interested participants and their Legally acceptable representative (LAR) will be administered the written informed consent. The participant will be screened and on fulfilling the inclusion and exclusion criteria will be enrolled into the study.

Socio demographic details will obtained from the participants. Baseline laboratory analysis which includes complete blood count, random blood sugar, liver function test, renal function test, urine analysis, ECG will be done for all the participants to screen for fitness. Urine pregnancy test will be done for women participants in the reproductive age group.

Positive and Negative Syndrome Scale (PANSS) will be administered to the participants.

Brief assessment of Cognition in Schizophrenia (BACS) will be administered in the following order i. List learning ii. Digit sequencing task iii. Token motor task iv. Verbal fluency: Category Instances, Controlled Oral Word Association Test v. Tower test vi. Symbol coding The study drug Tab. Prucalopride 1 mg (30 tablets) will be dispensed to the participant. They will be explained to take one tablet of 1 mg Prucalopride per oral in the morning. The participants will continue their antipsychotic regimen as per orders of their consultant and will continue to purchase their psychiatric medications as earlier. At the end of week 1, participants will be assessed for side effects via telephonic conversation.

At the end of 4 weeks, the participants will be scheduled for the assessments. Laboratory analysis, PANSS and BACS will be administered. Any side effects to the drug will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as schizophrenia by DSM 5 criteria using Structured Clinical Interview for DSM disorders
* Age between 18 to 55 years
* A minimum of one year of duration of illness
* Clinically stable with a stable therapeutic dose for at least 3 months prior to the recruitment
* Participants who can read and write English or Kannada

Exclusion Criteria:

* Participants who are acutely symptomatic and are uncooperative for assessments
* Co morbid with other psychiatric illness including mood disorders and substance use disorders except tobacco
* Participants already diagnosed with Intellectual Disability Disorder, head injury
* Participants administered MECT (modified electroconvulsive therapy)
* Participants with sensory impairments
* Use of Donepezil, Rivastigmine, Memantine, Benzodiazepines
* Participants already on prucalopride
* Participants with contraindications to prucalopride
* Diagnosed with gastrointestinal disorders like Ulcerative colitis, Crohn's disease, Intestinal ulcers
* Use of concomitant herbal remedies, alternative medicines
* Women who are pregnant or lactating
* Current history of suicidal ideation, intention or attempts

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2026-07-31 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale for Schizophrenia (PANSS )Score | PANSS scores measured at baseline and at the end of 4 weeks
  There will be change is PANSS score at the end of the study. The score is to assess symptoms. Lowest score is 30 and highest is 210.
Cognitive Functioning (List learning) | Baseline and and at the end of 4 weeks
  To study the change in the cognitive functioning as measured by list learning after intervention. Scores range between 0 and 30.
Cognitive Functioning (Digit sequencing task) | Baseline and and at the end of 4 weeks
  To study the change in the cognitive functioning as measured by Digit sequencing task after intervention, It ranges from 0 to 28 points
Cognitive Functioning (Token motor task) | Baseline and and at the end of 4 weeks
  To study the change in the cognitive functioning as measured by Token motor task after intervention. It ranges from 0 to 100 points,
Cognitive Functioning (Tower test) | Baseline and and at the end of 4 weeks
  To study the change in the cognitive functioning as measured by Tower test after intervention
Cognitive Functioning (Symbol coding) | Baseline and and at the end of 4 weeks
  To study the change in the cognitive functioning as measured by Symbol coding after intervention. It ranges from 0 to 22 points.

CONTACTS AND LOCATIONS:
Overall Officials: Vishwajit L Nimgaonkar, MD, PhD, Principal Investigator — University of Pittburgh
Locations (1):
- K S Hegde Medical Academy,, Mangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: One year after publication of this study.
Access Criteria: For individual participant data, meta-analysis.